CLINICAL TRIAL: NCT03291873
Title: Topography-Guided Customized PRK (Photorefractive Keratectomy) Versus Q-value Adjusted PRK in Correction of Myopia With or Without Astigmatism
Brief Title: Topography-Guided Customized PRK Versus Q-value Adjusted PRK in Correction of Myopia With or Without Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rania Elsayed Gad, Assisstant lecturer Faculty of Medicine Helwan University, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 900800700600500400300200100900
Record Dates: First submitted 2017-08-08; First posted 2017-09-25 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topography guided PRK in one eye (Active Comparator): Topography-guided (placido disk- based) using T-CAT Contoura treatment.
  Interventions: Procedure: PRK
- Q-value adjusted ( custom Q) PRK in the other eye (Active Comparator): The target Q will be estimated according to a nomogram considering the patient's age
  Interventions: Procedure: PRK

INTERVENTIONS:
Procedure: PRK — PRK using Alcon-Wavelight Excimer Laser EX 500

SUMMARY:
This study will include patients who will undergo PRK in both eyes, for each patient each eye will be randomly allocated to one of 2 procedures:

topography-guided ablation in one eye (group I) and Q-factor customized ablation in the other eye (group II).

Alcon/Wavelight Light Laser Technolo¬gie (GmbH, Erlangen, Germany) will be used for photoablation.

The wavelight Topolyzer (Wavelight AG, Erlan¬gen, Germany)and CSO Sirius scheimpflug camera combined with Placido corneal topography (CSO, Florence,Italy) will be used before and 1, 3 and 6 months after PRK. Refrac¬tive visual outcomes and corneal aberration changes will be compared between the two treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Myopia with up to -6.5 D with or without astigmatism up to -4.75 D

Exclusion Criteria:

* anterior segment abnormalities (ie, cataracts, corneal scarring)
* basement membrane disease
* history of recurrent corneal erosions
* Schirmer's test less than 5 mm
* established or forme fruste keratoconus
* macular or retinal disease
* current use of immunosuppressive therapy
* autoimmune disease
* pregnancy, and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
change in Postoperative spherical equivalent depending on manifest refraction after autorefractometer | 1 , 3 and 6 months postoperative
change in visual acuity using snellen chart | 1 , 3 and 6 months postoperative
change in corneal wavefront aberrations | 1 , 3 and 6 months postoperative
  assessed by topolyzer
change in Q value anterior at 6mm RMS, RMS of astigmatism, RMS of coma and RMS of spherical aberrations. Strehl ratio : Qvalue,RMS,strehl ratio by CSO Sirius scheimpflug | 1,3 and 6months
  by CSO Sirius scheimpflug
change in total RMS | 1,3 and 6months
  by CSO Sirius scheimpflug
change in strehl ratio | 1,3 and 6 months
  by CSO scheimpflug
change in Q value | 1,3 and 6 months
  assessed by topolyzer

SECONDARY OUTCOMES:
efficacy:ratio of postoperative decimal UDVA to preoperative decimal CDVA | 6 months
  ratio of postoperative decimal UDVA to preoperative decimal CDVA
contrast sensitivity | 6 months
  cambridge low contrast sensitivity
predictability | 6 months
  eyes within 1.0 D of emmetropia
safety:ratio of mean preoperative decimal CDVA to mean postoperative decimal CDVA | 6 months
  ratio of mean preoperative decimal CDVA to mean postoperative decimal CDVA
stability | 6 months
  change of more than 0.5D over

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Eyecare centre, Maadi, Cairo Governorate
  - Dar Al Oyun hospital, Giza

IPD SHARING:
Plan to Share IPD: Undecided